CLINICAL TRIAL: NCT04616781
Title: Effects of Ketone Ester on Brain Function and Alcohol Consumption in Alcohol Use Disorder
Brief Title: Ketone Ester Intervention in Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 844235; 4R00AA026892-02 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-11-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder
Keywords: Ester Keytone; MRI
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: The study is a randomized, 2-way placebo-controlled crossover trial in 20 non-treatment seeking individuals with AUD.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone ester with alcohol consumption (Active Comparator): Drink a single dose of ketone ester 1.9 kcal/kg, complete 1 hour MRI scan, drink an alcohol priming dose to produce a 0.03 g/dl breath alcohol concentration (BrAC) followed by a choice paradigm in which subjects receive 2 trays of 4 min-drinks each beverages Each min-drink would achieve 0.015 g/ld BrAC over a 1 hour period to achieve a max 0.1 g/dl BrAC.
  Interventions: Dietary Supplement: Ketone Ester "(R)-3-hydroxybutyl (R)-3-hydroxybutyrate"; Other: Alcohol drinks
- Isocaloric dextrose placebo drink with alcohol consumption (Placebo Comparator): Drink a single dose of Isocaloric dextrose placebo drink, complete 1 hour MRI scan, drink an alcohol priming dose to produce a 0.03 g/dl breath alcohol concentration (BrAC) followed by a choice paradigm in which subjects receive 2 trays of 4 min-drinks each beverages Each min-drink would achieve 0.015 g/ld BrAC over a 1 hour period to achieve a max 0.1 g/dl BrAC.
  Interventions: Drug: Isocaloric dextrose placebo; Other: Alcohol drinks

INTERVENTIONS:
Dietary Supplement: Ketone Ester "(R)-3-hydroxybutyl (R)-3-hydroxybutyrate" — nutritional ketone ester
  Other Names: Delta G
  Arms: Ketone ester with alcohol consumption
Drug: Isocaloric dextrose placebo — Drink indistinguishable from ketone ester
  Arms: Isocaloric dextrose placebo drink with alcohol consumption
Other: Alcohol drinks — drink an alcohol priming dose to produce a 0.03 g/dl breath alcohol concentration (BrAC) followed by a choice paradigm in which subjects receive 2 trays of 4 min-drinks each beverages Each min-drink would achieve 0.015 g/ld BrAC over a 1 hour period to achieve a max 0.1 g/dl BrAC.

SUMMARY:
The purpose of this research is to study how a nutritional ketone ester may effect brain function and alcohol consumption in regular alcohol users. The study will see how the brain responds, once after drinking the ketone ester and once after drinking a "placebo", which will look and taste the same as the ketone ester drink.

Metabolic ketosis induced by a ketogenic diet has been previously shown to elevate brain ketone bodies and reduce alcohol withdrawal symptoms in humans with AUD, and reduce alcohol consumption in alcohol-dependent rats. The study investigates whether metabolic ketosis induced by a one-dose nutritional ketone ester (KE) reduces brain reactivity to alcohol cues (fMRI), alcohol craving and alcohol consumption in humans with AUD, and if KE elevates ketone bodies using proton spectroscopy. This study uses a double blind, random ordered, 2-way crossover design in n=20 non-treatment seeking AUD who come in on two separate testing days: on one testing day the participants consume KE ((R)-3-hydroxybutyl (R)-3-hydroxybutyrate), and on another testing day a drink with isocaloric dextrose (DEXT), after which participants are scanned for 1H-MRS and fMRI and complete an alcohol consumption paradigm each day after scanning.

DETAILED DESCRIPTION:
This is a one month, prospective, double-blind, randomized, 2-way crossover design in n=20 non-treatment seeking AUD who come in for a screening day and two separate testing days: on one testing day the participants consume a drink with 1.9 kcal/kg of nutritional ketone ester (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (KE), and on another testing day a drink with isocaloric dextrose (DEXT), after which participants are scanned for 1H-MRS and fMRI (20 subjects are scanned twice; 40 scans in total) and complete an alcohol consumption paradigm each day after scanning (40 in total). Blood labs for ketone bodies, ghrelin and leptin will be drawn during the study visists.

The KE "(R)-3-hydroxybutyl (R)-3-hydroxybutyrate" is a safe, effective, and non-invasive way to increases ketone levels within 1 hr to concentrations similar to KD, and does not require a study IND. KE-induced ketone levels remain heightened for 4 hrs, and one dose of KE has shown to increase athletes' performances, improve mood, and cognitive and daily activity performance in Alzheimer's disease, and decrease ghrelin levels and subjective appetite in healthy volunteers. The latter finding is relevant to AUD, since ghrelin has been positively associated with alcohol craving and alcohol self-administration in AUD patients.

Before study participation, subjects are screened for psychiatric and medical problems, fasting glucose, urine drug screen, pregnancy test if female.

On each testing day, both before and 30 min after the drink, ketone bodies, leptin and ghrelin are measured in blood. After 15 minutes of KE, participants undergo a 1-hour MRI scan during which, after standard structural scans, the investigators measure ketone body metabolites using 1H-MRS, reactivity to alcohol cues using functional MRI, resting state MRI, cerebral blood flow using perfusion and brain iron measurements.

On each study visit, four blood draws will be analyzed for ketone bodies, ghrelin and leptin at KE intake (t0), 15 minutes after when the MRI starts (t15), 10 after the MRI is done and after the priming drink (t85), and then at 140, and 200 minutes after (i.e., t140 and t200).

Directly after MRI scanning, participants perform an alcohol self-administation "bar-lab" paradigm. Alcohol craving and alcohol effects will be measured before and during the alcohol self-administration. Participants will then be asked what they thought the study was about, and whether they thought the experimental drink influenced them in any way. After this, participants will be breathalyzed, and receive a meal.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years to 65 years old.
2. Willingness to provide signed, informed consent and commit to completing the procedures in the study
3. Meets DSM-5 criteria for AUD
4. Average weekly ethanol consumption of at least 15 standard drinks over the past month prior to consent (self-report)
5. Participants not seeking treatment for their AUD (self-report)
6. Alcohol specified as the preferred drug (self-report).
7. Women of child-bearing potential (i.e., who have not had a hysterectomy, bilateral oophorectomy, tubal ligation or is less than two years postmenopausal): must be non-lactating and practicing a reliable method of birth control, and have a negative urine pregnancy test prior to the initiation of the study and MRI procedures. Examples of medically acceptable methods for this protocol include: the birth control pill, intrauterine device (no copper IUD), injection of Depo-Provera, Norplant, contraceptive patch, contraceptive ring, double-barrier methods (such as condoms and diaphragm/spermicide), male partner sterilization, abstinence (and agreement to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence), and tubal ligation.

Exclusion Criteria:

1. Unwilling or unable to refrain from use, within 24 hours of MRI procedures, psychoactive medications or medication that may affect study results (e.g., analgesics containing narcotics, antibiotics, anti-inflammatory drugs).
2. Current DSM-5 diagnosis of a major psychiatric disorder (other than alcohol and nicotine use disorders, or substance use disorders that are mild/moderate) that required hospitalization, or that required daily medications for over 4 weeks in the past year (i.e., antidepressants; anticholinergics; antipsychotics; anxiolytics; lithium; psychotropic drugs not otherwise specified (nos) including herbal products (no drugs with psychomotor effects or with anxiolytics, stimulant, antipsychotic, or sedative properties); sedatives/hypnotics).
3. Urine drug screen positive for recent use of opioids, cocaine, or amphetamines on study visits (may be repeated once and if the result is negative on repeat it is not exclusionary).
4. A current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation that can impact brain function, the use of a ketone ester or the use of alcohol (e.g., epilepsy, diabetes, liver disease, kidney disease, kidney stones, chronic metabolic acidosis or a cardiomyopathy as determined by history and clinical exam).
5. Currently suffering from or with a history of stroke and/or stroke related spasticity.
6. History of seizures.
7. HIV positive, as the human immunodeficiency virus affects the brain.
8. Head trauma with loss of consciousness for more than 30 minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI. (self-report, medical history).
9. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head, fear of enclosed spaces, or other standard contraindication to MRI (self-report checklist).
10. Claustrophobia or other medical condition preventing subject from lying comfortably flat on his/her back for up to 2 hours in the MRI scanner (self-report).
11. BMI > 35, body girth greater than 52 inches and a head girth greater than 25 inches (imaging data acquisition is impaired with high-weight individuals).
12. Vision problems that cannot be corrected with glasses.
13. Judged by the principal investigator or his designee to be an unsuitable candidate for study participation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Determine the effects of ketone ester "R)-3-hydroxybutyl (R)-3-hydroxybutyrate" (KE) on alcohol consumption | 4 hours
  Compare the number of alcoholic drinks consumed in a "bar lab" paradigm after KE versus the Placebo drink
Determine the effect of KE on alcohol craving | 4 hours
  Compare the response to alcohol craving questionnaires after KE versus the Placebo drink
Determine the effect of KE on brain reactivity to alcohol cues | 2 hours
  Compare Brain reactivity to alcohol cues as measured with functional MRI after KE versus the Placebo drink

SECONDARY OUTCOMES:
Determine whether KE elevates brain ketone bodies using magnetic resonance spectroscopy | 2 hours
  Compare brain ketone levels after KE versus the Placebo drink
Determine whether ghrelin levels in blood covary with alcohol craving and consumption | 4 hours
  Correlate blood ghrelin levels with alcohol craving questionnaire scores and number of alcoholic drinks consumed, at KE versus Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Corinde E Wiers, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States